CLINICAL TRIAL: NCT04269356
Title: Pharmacokinetics and Metabolism of a Single Dose of [14C] BMS-986256 in Healthy Male Participants
Brief Title: Study to Assess the Way the Body Absorbs, Distributes, Breaks Down and Eliminates Radioactive BMS-986256 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM026-023
Record Dates: First submitted 2020-02-12; First posted 2020-02-13 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Magnesium Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986256 (Experimental)
  Interventions: Drug: BMS-986256; Drug: Milk of magnesia

INTERVENTIONS:
Drug: BMS-986256 — Specified dose on specified days
Drug: Milk of magnesia — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the way the body absorbs, distributes, breaks down and eliminates radioactive BMS-986856 in healthy males.

DETAILED DESCRIPTION:
Recruitment temporarily on hold due to COVID-19.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participants, as determined by no clinically significant deviations from normal in medical history, physical examination abnormalities that would compromise the ability to participate, complete, and/or interpret the results of the study, 12-lead electrocardiograms (ECGs), vital signs, and clinical laboratory results.
* Males must agree to follow specific methods of contraception, if applicable, while participating in the trial

Exclusion Criteria:

* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study
* History of any significant drug and/or food allergies

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of [14C] BMS-986256 | Up to 49 days
Time to attain maximum observed plasma concentration (Tmax) of [14C] BMS-986256 | Up to 49 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC (0-T)) of [14C] BMS-986256 | Up to 49 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 49 days
Incidence of Serious Adverse Events (SAEs) | Up to 49 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 49 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 49 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 49 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 49 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 49 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 49 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 49 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters | Up to 49 days
Incidence of clinically significant changes in physical examination findings | Up to 49 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance - Clinical Pharmacology Services - Madison, Madison, Wisconsin, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm